CLINICAL TRIAL: NCT06636474
Title: Evaluation of the Supported Housing System for the Inclusion of People Suffering From Mental Disorders
Acronym: EVA-DLAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D20-P007
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: All patients benefiting from a DLAI and suffering from psychiatric disorders, monitored in sector 75G08-09 of the Saint-Maurice hospitals, and sectors 75G19, 75G20-21, 75G25, 75G26 of the GHU Paris.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with mental disorders (Other): administration of standardized questionnaires and scales, upon entering the research, then annually, and finally upon leaving the research
  Interventions: Other: patients with mental disorders

INTERVENTIONS:
Other: patients with mental disorders — administration of standardized questionnaires and scales, upon entering the research, then annually, and finally upon leaving the research

SUMMARY:
Access to housing, in the current context of extreme tension in the rental housing market in Paris and throughout the Ile-de-France region, is proving to be extremely complex for people with mental health problems.National and international scientific studies have quantified the problem of homelessness and precarious or inappropriate housing among patients suffering from psychiatric disorders, and show the impact of housing problems on the consumption of psychiatric care.The DÉLAI's mission is to facilitate access to housing for people enrolled in a psychiatric care pathway, with teams from the psychiatric sectors

DETAILED DESCRIPTION:
* Written and oral information provided to the patient by the patient's referring psychiatrist (Investigator of one of the five recruiting sites) during a regular consultation appointment.
* Initial assessment (V inclusion): reminder of the information concerning the research, collection of consent, collection of sociodemographic data, and standardized assessment scales (quality of life, clinical state, level of functioning) + standardized semi-structured interview for the diagnosis of psychiatric disorders + completion by the referring psychiatrist of the data corresponding to the patient's care pathway.
* Then follow-up visit at an annual rate (V1 ... VX), and DLAI exit assessment (V exit) as soon as the patient stops benefiting from the DLAI.

ELIGIBILITY:
Inclusion Criteria:

patient followed for a psychiatric disorder patient benefiting from a DLAI

Exclusion Criteria:

patient not followed for psychiatric disorder patient who refused to participate in the research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2030-07-27 (Estimated); Study Completion 2030-12-27 (Estimated)

PRIMARY OUTCOMES:
improvement of quality of life | one year
  World Health Organization Quality of Life-26,26-item self-assessment questionnaire for assessing quality of life covering four major dimensions: physical health, mental health, social relationships and environment
improvement of quality of life | one year
  quality of life rating scale (each item is rated from 0 to 6, giving a total score out of 42 points), assessing interpersonal relationships (relationships with close acquaintances and social initiatives), social status, intrapsychic functioning (degree of motivation, anhedonia and capacity for empathy) and regular activities.

SECONDARY OUTCOMES:
clinical condition | one year
  Mini International Neuropsychiatric Interview : structured diagnostic interview, relatively short in duration, exploring in a standardized way the main psychiatric disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France